CLINICAL TRIAL: NCT02430246
Title: The Association Between the Transfer of Lactobacilli From the Gastrointestinal Tract to the Vagina and the Prevention / Eradication of Abnormal Vaginal Flora in High Risk Pregnancies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After completing the part of assessing lactobacilli transfer, it was decided not to proceed further with the masked part of the study.
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, enav yefet, MD/PhD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0096-13
Record Dates: First submitted 2015-04-20; First posted 2015-04-30 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Pregnancy
MeSH Terms: interventions — methenamine hippurate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Primary prevention - Urex Plus (Experimental): Patients with Normal vaginal flora in the experimental arm will be treated with UREX PLUS
  Interventions: Dietary Supplement: Urex Plus
- Primary prevention - Placebo (Placebo Comparator): Patients with Normal vaginal flora in the Placebo arm will be treated with a capsule without active ingredient
  Interventions: Other: Placebo
- Secondary prevention - Urex Plus (Experimental): Patients with abnormal vaginal flora in the experimental arm will be treated with antibiotic (either clindamycin, metronidazole or both if one was not effective), Once AVF/BV was eradicated, the patient will be given UREX PLUS
  Interventions: Dietary Supplement: Urex Plus
- Secondary prevention - Placebo (Placebo Comparator): Patients with abnormal vaginal flora in the Placebo arm will be treated with antibiotic (either clindamycin, metronidazole or both if one was not effective), Once AVF/BV was eradicated, the patient will be given placebo without active ingredient
  Interventions: Other: Placebo
- Eradication - Urex Plus (Experimental): Patients with persistent abnormal vaginal flora following treatment with clindamycin and metronidazole in the experimental arm will be treated with UREX PLUS
  Interventions: Dietary Supplement: Urex Plus
- Eradication - Placebo (Placebo Comparator): Patients with persistent abnormal vaginal flora following treatment with clindamycin and metronidazole in the placebo arm will be treated with placebo without active ingredient
  Interventions: Other: Placebo
- Lactobacilli transfer - probiotic capsule (Other): Patients with Normal vaginal flora will be treated with a probotic capsule containing L. rhamnosus GR-1and L. reuteri RC-14 for two months afterwhich they will receive no treatment for additional two months. Lactobacili colonization in the vaginal flora will be tested
  Interventions: Dietary Supplement: Probotic capsule containing L. rhamnosus GR-1and L. reuteri RC-14
- Lactobacilli transfer - probiotic capsule after 2 months (Other): Patients with Normal vaginal flora will be followed for two months without intervention afterwhich they will receive a probotic capsule containing L. rhamnosus GR-1and L. reuteri RC-14 for two months. Lactobacili colonization in the vaginal flora will be tested.
  Interventions: Dietary Supplement: Probotic capsule containing L. rhamnosus GR-1and L. reuteri RC-14

INTERVENTIONS:
Dietary Supplement: Urex Plus — Probiotic
  Arms: Eradication - Urex Plus; Primary prevention - Urex Plus; Secondary prevention - Urex Plus
Other: Placebo — capsule without active ingredient
  Arms: Eradication - Placebo; Primary prevention - Placebo; Secondary prevention - Placebo
Dietary Supplement: Probotic capsule containing L. rhamnosus GR-1and L. reuteri RC-14
  Arms: Lactobacilli transfer - probiotic capsule; Lactobacilli transfer - probiotic capsule after 2 months

SUMMARY:
Pregnant women at high risk for preterm labor from at least 13 weeks of gestation will be tested to detect abnormal vaginal flora (AVF) or its severe form - bacterial vaginosis (BV) by taking vaginal smear. Treatment will be given according to the results.

DETAILED DESCRIPTION:
Pregnant women at high risk for preterm labor from at least 13 weeks of gestation will be tested to detect AVF/BV by taking vaginal smear. Diagnosis will be according to the Nugent score criteria. Treatment will be given according to the results:

Patient with a positive smear for AVF- patients tested positive will be treated with either clindamycin or metronidazole. Following treatment another smear will be taken according to which the patients will be divided into 2 research groups: (1) Assessing the effectiveness of probiotic formula to prevent AVF re-infection (secondary infection) - this group includes patients with normal vaginal flora following antibiotic administration. (2) Assessing the effectiveness of probiotic formula to eradicate AVF - this group includes patients with persistent AVF following antibiotic administration (first and second line). In each group the patients will be divided into a research group which will receive the probiotic formula UREX PLUS (containing L. rhamnosus GR-1and L. reuteri RC-14) and a control group which will receive a placebo twice a day until 36.6 weeks of gestation.

Patient with a negative smear for AVF - in those patients the effectiveness of probiotic formula will be tested for primary prevention. These patients will be divided into a research group which will receive the probiotic formula UREX PLUS and a control group which will receive a placebo twice a day until 36.6 weeks of gestation.

Finally, the colonization of lactobacilli in the vaginal flora will be examined by dividing patients with normal vaginal flora into one group receiving a probiotic capsule containing L. rhamnosus GR-1 and L. reuteri RC-14 twice a day for 2 months and a second group without intervention. After two months the group receiving probiotic capsule will receive no treatment and the second group will receive probiotic capsule containing L. rhamnosus GR-1and L. reuteri RC-14 twice a day for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women from at least 13 weeks of gestation with a risk factor for preterm labor

Exclusion Criteria:

* Women with preterm premature rupture of the membranes
* Immunocompromised women
* Planned elective preterm birth for reasons other than preterm premature rupture of membranes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03-14 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
The amount of lactobacilli in the vaginal | once a month until week 36.6 of labor
  Lactobacilli culture will be made from a vaginal specimen. The pattern of bacterial growth will be used for a semi-quantitative interpretation in a scale of 0-no vaginal colonization to 4-substantial colonization.
The rate of women with normal vaginal flora at enrollment, who developed AVF/BV during the study period | From date of randomization until the date of first documented episode or until delivery (around 4 months)
The rate of women with AVF/BV at enrollment whose infection was eradicated following antibiotics, who developed AVF/BV during the study period | From date of randomization until the date of first documented episode or until delivery (around 4 months)
The rate of women with AVF/BV at enrollment whose infection was not eradicated following antibiotics, who restored the normal vaginal flora during the study period | Until delivery (around 4 months)

SECONDARY OUTCOMES:
Duration of time from the beginning of the study until an episode of AVF/BV | From date of randomization until the date of first documented episode or until delivery (around 4 months)
The number of episodes of BV/AVF during pregnancy | Until delivery (around 4 months)
The rate of women, who suffer from obstetrical outcomes(preterm labor, intrauterine growth restriction, preterm premature rupture of membranes, chorioamnionitis, post-partum fever, post-partum endometritis, neonatal sepsis and neonatal complications) | Until delivery (around 4 months)
The rate and type of adverse effects in the probiotic versus placebo groups | Until delivery (around 4 months)
Number of urinary tract infections during the study period | Until delivery (around 4 months)

CONTACTS AND LOCATIONS:
Overall Officials: ENAV YEFET, MD/PhD, Principal Investigator — HaEmek Medical Center , Afula
Locations (1):
- HaEmek Medical Center, Afula, Israel